CLINICAL TRIAL: NCT05155371
Title: Titration of Intraoperative Positive End-expiratory Pressure to Optimize Gas Exchange in Patients Undergoing Robotic Assisted Laparoscopic Prostatectomy
Brief Title: Titration of Intraoperative PEEP in Patients Undergoing Robotic Assisted Laparoscopic Prostatectomy
Acronym: TIPPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Department of Anesthesiology, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: PEEP Titration of RALP
Record Dates: First submitted 2021-11-18; First posted 2021-12-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Positive End Expiratory Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Positive End-expiratory Pressure obtained with Titration of Fraction of Inspiratory Oxygen (Experimental): Obtained Optimal Positive End-expiratory Pressure obtained with Titration of Fraction of Inspiratory Oxygen and sustained the PEEP intraoperatively
  Interventions: Other: Titration of Optimal Positive End-expiratory Pressure
- Optimal Positive End-expiratory Pressure obtained with electrical impedance tomography (Experimental): Obtained Optimal Positive End-expiratory Pressure obtained with EIT and sustained the PEEP intraoperatively
  Interventions: Other: Titration of Optimal Positive End-expiratory Pressure

INTERVENTIONS:
Other: Titration of Optimal Positive End-expiratory Pressure — Titration of Optimal Positive End-expiratory Pressure with two different methods

SUMMARY:
Optimal intraoperative positive end expiratory pressure (PEEP) improves the outcome. Optimal PEEP is not only very different among individuals, but each individual's optimal PEEP is affected by positioning, muscle paralysis, and several other factors. Several techniques have been used to determine the optimal PEEP. For example, electrical impedance tomography(EIT)can be performed at the bedside.However, the application of this technique requires special training, increases the workload of the care team, and the cost-efficiencyof this procedure remains to be determined.We hypothesized that optimal PEEP could be obtained by titration of intraoperative PEEP levels and FiO2with SpO2 guidance. Our secondary hypothesis was that maintenance of intraoperative optimal PEEP derived via this method improves intraoperative oxygenation and reduces the incidence of postoperative hypoxemia.We tested our hypothesis in patients undergoing robotic-assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
Lung-protective ventilation strategies are recommended for patients under mechanical ventilation with intermediate-risk and high-risk in order to minimize lung injury and respiratory complications of critically ill patients associated with mechanical ventilation , such as atelectasis and pneumonia. Low tidal volume (TV) had been proven protective . However, there is no consensus on what the optimal positive end expiatory pressure (PEEP) is for patients with healthy lungs undergoing general anesthesia, particularly for those who are undergoing abdominal surgery. A recent study showed that electrical impedance tomography (EIT) could be used to identify optimal PEEP, where both lungs collapse, hyper-insufflation is minimized, and the variation of optimal PEEP in patients with healthy lungs undergoing abdominal surgery is profound.Therefore, a fixed PEEP applied to all patients surely over-PEEP some and under-PEEP others. This study also demonstrates that maintaining the optimal PEEP intra-operatively not only improves intra-operative oxygenation but also reduces the incidence and severity of atelectasis post-operatively . Even though this study focuses on the improvement of physiology rather than the outcome, the benefit of intra-operative optimal PEEP is sustained for at least for one-hour post extubation. Therefore, optimized intra-operative PEEP could potentially have a positive impact onoutcomes. However, the cost-effectiveness of EIT used intraoperatively as routine practice still needs to be determined. Development of new methods which can be used intraoperatively and arecost-effective and user-friendly is an unmet demand.

Recently, Ferrando et al conducted a study in which the authors used minimal FiO2 to maintain clinically acceptable arterial blood O2 saturation by titrating PEEP. Even though this study was not randomized and sample size was insufficient to demonstrate improved outcomes, it clearly demonstrated its feasibility and safety. We hypothesize that titration of intraoperative PEEP using minimal FiO2 while maintaining clinically acceptable O2 saturation allows clinicians to identify the optimal PEEP. We will test this hypothesis on patients undegoing RALP. We chose this population because these patients have increased number of postoperative complications . Additionally, physicians are prone to using suboptimal ventilation strategies such as inappropriate tidal volumes and intraoperative PEEP in this population; therefore these patients are more likely to achieve maximal benefit with optimized intra-operative PEEP.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 years or older
* scheduled for elective robotic-assisted laparoscopic prostatectomy(RALP)
* ASA physical status of I-III

Exclusion Criteria:

* acute or chronic respiratory disorders
* pulmonary hypertension
* neuromuscular disease
* preoperative SpO2<95% on room air

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
The difference of optimal PEEP titrated by two methods | within 30 minutes after trachea intubation
  Titration result of the two groups

SECONDARY OUTCOMES:
Difference of intraoperative PaO2/FiO2 between the two groups | 30,60,120 minutes after finishing PEEP titration
  intraoperative PaO2/FiO2 between the two groups
Difference of intraoperative driving pressure, dynamic compliance between the two groups | 30,60,120 minutes after finishing PEEP titration
  Difference of intraoperative driving pressure, dynamic compliance between the two groups
Difference of lung regional ventilation between the two groups | 5 minutes after trachea extubation
  lung regional ventilation recorded by EIT
Post operation hypoxemia in PACU. | within 30 minutes after trachea extubation
  Postoperative hypoxemia was defined as postoperative hypoxemia if SpO2<92%was detected in room air within 30 min after extubation in the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Study Chair — Department of Anesthesiology, Fudan University Shanghai Cancer Center; Department of Oncology, Shanghai Medical College, Fudan University
Locations (2):
- China (2):
  - 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No